CLINICAL TRIAL: NCT03189394
Title: A Randomized Trial to Prevent HIV Among Gay Couples
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Francisco State University (Other)
Collaborators: University of California, San Francisco (Other); University of Colorado, Denver (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20419000
Record Dates: First submitted 2017-04-05; First posted 2017-06-16 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: HIV Infections
Keywords: HIV; gay couples; relationships; dyads
MeSH Terms: conditions — HIV Infections | interventions — Men's Health

STUDY DESIGN:
Intervention Model Description: On completion of the baseline survey and testing, couples will be randomized to one of the three arms of the study (PRIDE, ePRIDE, or Men's Health). Couples will be randomized in blocks with the block size randomly permuted via a SAS computer program based on a pseudo-random number generator. Each arm of the intervention will begin on the same date and run for two weeks. Couples randomized to ePRIDE will be sent a link on the same day that PRIDE and Men's Health sessions are scheduled and will have two weeks to complete the program.
Who Masked: Participant
Masking Description: Participants will be aware that there are online and in-person aspects of the study as seen in the consent form, but will be randomized to a group and unaware of which arm they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRIDE (Experimental): The in-person experimental condition, PRIDE, consists of in-person intervention activities that are scheduled over two Saturdays, back to back, approximately 3 hours each (6 hours total). This intervention consists of relationship-focused activities for couples to take part in together, focusing on relationship communication, dynamics, and sexual agreements.
  Interventions: Behavioral: PRIDE
- ePRIDE (Experimental): ePRIDE is an online adaptation of the experimental condition, PRIDE, and consists of online intervention activities that are scheduled to be completed over two weeks, lasting approximately 6 hours total. This intervention consists of relationship-focused activities for couples to take part in together, focusing on relationship communication, dynamics, and sexual agreements, and is designed for couples to take together sitting side by side.
  Interventions: Behavioral: ePRIDE
- Men's Health (Active Comparator): Men's Health is the active comparator group. Participants in this group go through in-person intervention days, scheduled on Saturdays back to back, but differ from the PRIDE arm because this intervention does not focus on relationship dynamics. Instead, these two Saturday intervention days focus on general men's health, including heart health, cancer, and STDs.
  Interventions: Behavioral: Men's Health

INTERVENTIONS:
Behavioral: PRIDE — A couples curriculum that is relationship-focused and in-person, aimed at helping to reduce the odds of a composite HIV risk variable among gay couples.
  Arms: PRIDE
Behavioral: ePRIDE — A couples curriculum that is relationship-focused and online, aimed at helping to reduce the odds of a composite HIV risk variable among gay couples.
  Arms: ePRIDE
Behavioral: Men's Health — A men's health curriculum that is individualized and in-person, aimed at helping participants to focus on gay men's health.
  Arms: Men's Health

SUMMARY:
The proposed study is a randomized controlled intervention to reduce sexual risk for HIV among HIV-negative concordant and HIV discordant gay couples. There are three arms of the study: 1) the in-person experimental condition, PRIDE, 2) the online adaptation of the experimental condition, ePRIDE, and 3) the time- and attention-matched in-person control condition, Men's Health. Participants (N = 300 couples) will be randomized equally into one of the three study conditions and assessed via surveys at baseline and at 3-, 6- and 9-months after completion of the intervention sessions.

DETAILED DESCRIPTION:
Participants (N = 300 couples) will be randomized equally into one of the three study conditions and assessed via surveys at baseline and at 3-, 6- and 9-months after completion of the intervention sessions. All participants will complete a baseline survey, administered a fluid (swab) OraQuick HIV test, administered a viral load (VL) or PrEP adherence dry blood spot test using the HemaSpot collection device they will be randomized to one of three intervention arms, and then follow-up surveys will measure short and long term impact of the intervention at 3, 6, and 9 months.

They will first be provided with a brief overview of the study focusing on the goals of the study, randomization, participation details and timeline, and if they wish to proceed, will then be screened for eligibility. Our goal will be to screen and baseline cohorts of 30 couples (10 couples for each arm of the intervention) within a 6-week window (recruitment will be on-going).

Eligible couples will be scheduled to come into the study offices to complete a baseline survey. On arrival, couples will be informed in detail about the study and what their participation entails. Study staff will answer any outstanding questions, informed consent will be obtained, the participants will be given a fluid (swab) OraQuick rapid HIV test in a private CREGS office with HIV counseling-certified staff, then will give a DBS specimen for testing either viral load for HIV-positive participants or PrEP levels for HIV-negative participants. For consented and eligible participants, the baseline survey will then be administered and the baseline online survey will be administered on study computers.

On completion of the baseline survey and testing, couples will be randomized to one of the three arms of the study (PRIDE, ePRIDE, or Men's Health). Couples will be randomized in blocks with the block size randomly permuted via a SAS computer program based on a pseudo-random number generator. Each arm of the intervention will begin on the same date and run for two weeks. Couples randomized to ePRIDE will be sent a link on the same day that PRIDE and Men's Health sessions are scheduled and will have two weeks to complete the program. Access to ePRIDE will be deactivated at the end of two weeks.

Participants who have a positive test result for HIV during the baseline visit will be given their results by HIV counseling-certified staff and referred for free confirmatory testing at our nearby partner, Alliance Health Project clinic, where they will also receive clinical care and support services. If the newly HIV-positive person is in a relationship with a confirmed HIV-positive partner, they will be considered ineligible. If the partner is HIV-negative, they will be eligible to participate in the study.

Short and long term impact of the intervention will be measured at 3-, 6- and 9-months post completion of the intervention. Follow-up surveys for all three arms will be administered online in-person at the downtown CREGS offices. Couples will be sent a link to the survey with a unique identification number and password and will have 7 days to complete each survey; reminders will be sent every two days contacted and scheduled to come in together to complete follow-up surveys on provided computers. Couples who take fail to come in and complete follow-ups longer than 7 days will be flagged so differential outcomes can be assessed as needed and their link to the survey will be disabled after 14 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* speak English
* live in the San Francisco Bay Area
* have knowledge of their own and their partner's serostatus
* are in a concordant HIV-negative or discordant relationship
* at least one partner has had condomless anal sex (CAS) in the last three months
* identify as biologically male and not transgender
* in a committed relationship (defined as two men who are committed to each other above anyone else and have had sex with each other) with their primary male partner (who they will participate in the study with) for at least 3 months.

Exclusion Criteria:

* under 18
* do not speak English
* do not live in the San Francisco Bay Area
* do not know their own or their partner's HIV status
* are in a relationship where both partners are HIV positive, neither partner reports CAS in the last three months
* identifies as transgender
* is of female sex
* not in a current committed relationship for at least 3 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as biologically male and not transgender.
Enrollment: 600 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Composite Risk for HIV (CR-HIV) | 9 months (baseline, 3, 6, and 9 month followups)
  The primary outcome variable will be a binary indicator of any HIV-risk (no vs. yes) in the past three months at baseline, 3, months, 6 months, and 9 months--based on a composite of self-reported sexual risk behavior (defined as CAS with a discordant or unknown HIV status partner as well as HIV-positive partner's ART interruption (defined as missing all ART doses over a 4-day period in the past three months 70) and suppressed viral load. We will rely on self-reports of viral load because sexual risk behavior is based on one's perception of one's own or the partners' viral load. Regular viral load tests will be emphasized in PRIDE and ePRIDE to encourage participants to be proactive about their lab work. Baseline, 3 months, 6 months, and 9 months will be assessed for change over time past the date of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Hoff, PhD, Principal Investigator — CREGS, San Francisco State University
Locations (1):
- Center for Research and Education on Gender and Sexuaity (CREGS) At San Francisco State University, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No